CLINICAL TRIAL: NCT01516138
Title: Myocardial Protection of Glucose - Insulin - Potassium in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Benefits of GIK in Cardiac Surgery Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJcuiqin_2012
Record Dates: First submitted 2012-01-08; First posted 2012-01-24 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-07

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
Keywords: Glucose-insulin-potassium; Cardiac surgery
MeSH Terms: interventions — glucose-insulin-potassium cardioplegic solution; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GIK (Active Comparator): glucose-insulin-potassium (GIK) consists of 20% glucose (200 g/L), 66.7 U/L regular insulin and 80 mmol/L potassium chloride (KCl).
  Interventions: Drug: GIK
- Control (Placebo Comparator): 6.12 g/L sodium acetate, 5.85 g/L sodium chloride, 0.3 g/L potassium chloride and 0.33 g/L calcium chloride
  Interventions: Drug: Control

INTERVENTIONS:
Drug: GIK — Intravenous solution was started at about 10 minutes before general anesthesia, running at a rate of 1 mL/kg/h for 12.5 hours.
  Other Names: Glucose-insulin-potassium
  Arms: GIK
Drug: Control — Intravenous solution was started at about 10 minutes before general anesthesia, running at a rate of 1 mL/kg/h for 12.5 hours.
  Other Names: Balanced salt solution
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effects of modified glucose - insulin - potassium (GIK) therapy in cardiac surgery patients undergoing cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is a necessary technique to maintain the circulation during cardiac surgery. But CPB itself is associated with a series of problems of organs, such as hyperglycemia induced by neuroendocrine stress. The research showed that hyperglycemia induced by stress would cause a worsened hospital outcome for patients undergoing cardiac surgery. Intraoperative and postoperative glucose control is beneficial for patients.

It has been for more than 40 year since the first application of glucose - insulin - potassium (GIK) in cardiac surgery but the clinical application of GIK shows controversial results. The beginning time of application and the ratio of glucose and insulin may be the key reasons for the controversy. In our pilot trial of 40 valve replacement cases, we found that perioperative treatment of GIK with an insulin-glucose ratio of 1:3 showed beneficial effects during heart surgery. Therefore, the investigators are planning to continue to test this modified GIK regimen for more heart surgery patients and determine whether GIK may have cardioprotective effects on patients undergoing CPB surgery.

Myocardial biopsies for biological mechanism analysis will be performed prior to CPB, 15 min after aortic cross clamp application and 15 min after reperfusion only in a small cohort. Myocardial biopsies will be snap frozen or fixed.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age
* Elective cardiac surgery with first time cardiopulmonary bypass
* Left ventricular ejection fraction(LVEF) ≥ 30%
* Informed agreement signed

Exclusion Criteria:

* Previous cardiac surgery
* Emergent surgery
* Cardiac surgery without the use of cardiopulmonary bypass
* Diabetes mellitus
* Severe renal insufficiency
* Severe respiratory insufficiency
* Serious preoperative illness (sepsis, active infection or active malignancy requiring treatment)
* Pregnant woman or positive pregnancy test
* History of drug abuse
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion
* Enrollment in another clinical study
* Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants of the major adverse cardiac events | Stay in hospital
  The composite of major adverse cardiac events included acute myocardial infarction, cardiac arrest with successful resuscitation, low cardiac output syndrome, congestive heart failure, arrhythmia and all-cause death.

SECONDARY OUTCOMES:
mortality | until the study ends
Length of stay in intensive care unit and hospital | Stay in intensive care unit and hospital
  Length of stay in intensive care unit and hospital
Number of patients of postoperative complications | Stay in hospital
  Postoperative complications included prolonged ventilation, the use of inotropes, sepsis/infection, renal complications, stroke and reoperation.

OTHER OUTCOMES:
Left ventricular ejection fraction (LVEF) | 24h after operation and before discharge
Creatine kinase-myocardial bands (CK-MB) | during 48 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, MD,PhD, Study Chair — Deparment of cardiovascular surgery, XiJing hospital, Fourth Military Medical University; Qin Cui, MD,PhD, Principal Investigator — Deparment of cardiovascular surgery,XiJing hospital,Fourth Military Medical University; Jia Li, MD,PhD, Principal Investigator — Deparment of Physiology, Fourth Military Medical University; Feng Gao, MD,PhD, Principal Investigator — Deparment of Physiology, Fourth Military Medical University; Kun Zhao, MD, Principal Investigator — Deparment of cardiovascular surgery, XiJing hospital,Fourth Military Medical University; Shiqiang Yu, MD,PhD, Principal Investigator — Deparment of cardiovascular surgery, XiJing hospital, Fourth Military Medical University
Locations (1):
- Deparment of Cardiovascular surgery,Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zhao K, Zhang Y, Li J, Cui Q, Zhao R, Chen W, Liu J, Zhao B, Wan Y, Ma XL, Yu S, Yi D, Gao F. Modified Glucose-Insulin-Potassium Regimen Provides Cardioprotection With Improved Tissue Perfusion in Patients Undergoing Cardiopulmonary Bypass Surgery. J Am Heart Assoc. 2020 Mar 17;9(6):e012376. doi: 10.1161/JAHA.119.012376. Epub 2020 Mar 10. PMID 32151220